CLINICAL TRIAL: NCT02574455
Title: An International, Multi-Center, Open-Label, Randomized, Phase III Trial of Sacituzumab Govitecan Versus Treatment of Physician Choice in Patients With Metastatic Triple-Negative Breast Cancer Who Received at Least Two Prior Treatments
Brief Title: Trial of Sacituzumab Govitecan in Participants With Refractory/Relapsed Metastatic Triple-Negative Breast Cancer (TNBC)
Acronym: ASCENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-05; 2017-003019-21 (EudraCT Number)
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan (Experimental): Participants will receive sacituzumab govitecan on Days 1 and 8 of a 21-day treatment cycle for up to 29.6 months. Participants will continue treatment until progression of disease requiring treatment discontinuation or occurrence of unacceptable adverse events (AEs).
  Interventions: Drug: Sacituzumab govitecan
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive TPC (ie, eribulin, capecitabine, gemcitabine, or vinorelbine), administered as a single-agent regimen that is selected by the investigator before participant randomization. Participants will continue treatment until progression of disease requiring treatment discontinuation or occurrence of unacceptable AEs.
  Interventions: Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Sacituzumab govitecan — 10 mg/kg administered as a slow intravenous (IV) infusion either by gravity or with an infusion pump. Infusion rate for the first 15 minutes will start with 50 mg/hour or less with a subsequent infusion of 100 to 200 mg/hour up to a maximum recommended rate (advanced every 15 to 30 minutes) of 500 mg/hour with a subsequent infusion of 1000 mg/hour.
  Other Names: IMMU-132; Trodelvy®
  Arms: Sacituzumab Govitecan
Drug: Eribulin — Administered IV over 2 to 5 minutes at a dose 1.4 mg/m^2 at North American sites and 1.23 mg/m^2 at European sites on Days 1 and 8 of a 21-day cycle for up to 15.3 months. Lower doses will be administered on the same schedule to participants with moderate hepatic impairment (ie, Child-Pugh B; 0.7 mg/m^2 and 0.67 mg/m^2 for North American and European sites, respectively).
  Other Names: Halaven
  Arms: Treatment of Physician's Choice (TPC)
Drug: Capecitabine — 1000 to 1250 mg/m^2 will be administered in a 21-day cycle, with capecitabine administered orally twice daily for 2 weeks followed by 1-week rest period for up to 10.6 months.
  Other Names: Xeloda
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — 800 to 1200 mg/m^2 will be administered IV over 30 minutes on Days 1, 8, and 15 of a 28-day cycle for up to 8.1 months.
  Other Names: Gemzar
  Arms: Treatment of Physician's Choice (TPC)
Drug: Vinorelbine — 25 mg/m^2 will be administered as a weekly IV injection over 6-10 minutes for up to 11.5 months. Vinorelbine will not be allowed as TPC for any participant with Grade 2 neuropathy.
  Other Names: Navelbine
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The primary objective of this study is to compare the efficacy of sacituzumab govitecan to the treatment of physician's choice (TPC) as measured by independently-reviewed Independent Review Committee (IRC) progression-free survival (PFS) in participants with locally advanced or metastatic triple-negative breast cancer (TNBC) previously treated with at least two systemic chemotherapy regimens for unresectable, locally advanced or metastatic disease, and without brain metastasis at baseline.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed TNBC based on the most recent analyzed biopsy or other pathology specimen. Triple negative is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PR) and negative for human epidermal growth factor receptor 2 (HER2) by in-situ hybridization.
* Refractory to or relapsed after at least two prior standard therapeutic regimens for advanced/metastatic TNBC.
* Prior exposure to a taxane in localized or advanced/metastatic setting.
* Eligible for one of the chemotherapy options listed as TPC (eribulin, capecitabine, gemcitabine, or vinorelbine) as per investigator assessment.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Bone-only disease is not permitted.
* At least 2 weeks beyond prior anti-cancer treatment (chemotherapy, endocrine therapy, radiotherapy, and/or major surgery), and recovered from all acute toxicities to Grade 1 or less (except alopecia and peripheral neuropathy).
* At least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids < 20 mg prednisone or equivalent daily are permitted provided the dose is stable for 4 weeks).
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, absolute neutrophil count (ANC) > 1,500 per mm^3, platelets > 100,000 per mm^3).
* Adequate renal and hepatic function (creatinine clearance [CrCL] > 60 mL/min, bilirubin ≤ 1.5 institutional upper limit of normal [IULN], aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≤ 2.5 x IULN or ≤ 5 x IULN if known liver metastases and serum albumin ≥3 g/dL).
* Recovered from all toxicities to Grade 1 or less by National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) v4.03 (except alopecia or peripheral neuropathy that may be Grade 2 or less) at the time of randomization. Participants with Grade 2 neuropathy are eligible but may not receive vinorelbine as TPC.
* Participants with treated, non-progressive brain metastases, off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks can be enrolled in the trial.

Key Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential or fertile men unwilling to use effective contraception during study and up to three months after treatment discontinuation in women of child-bearing potential and six months in males post last study drug.
* Participants with Gilbert's disease.
* Participants with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while participants with other prior malignancies must have had at least a 3-year disease-free interval.
* Participants known to be human immunodeficiency (HIV) positive, hepatitis B positive, or hepatitis C positive.
* Infection requiring antibiotic use within one week of randomization.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (224):
- United States (179):
  - Southern Cancer Center, 29653 Anchor Cross Blvd, Daphne, Alabama
  - Souther Cancer Center, 3719 Dauphin St., 5 Floor, Mobile, Alabama
  - Southern Cancer Center, 3 Mobile Infirmary Circle, Mobile, Alabama
  - Southern Cancer Center, 6701 Airport Blvd., Bldg B, Terace Level, Mobile, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - UCLA Jonsson Comprehensive Cancer Center, 1411 S. Garfield Ave Suite 200, Alhambra, California
  - UCLA Jonsson Comprehensive Cancer Center, 201. S. Buena Vista St Suite 200, Burbank, California
  - UCLA Jonsson Comprehensive Cancer Center, Laguna Hills, California
  - UCLA Jonsson Comprehensive Cancer Center, 200 UCLA Medical Plaza, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, 625 South Fair Oaks Avenue Suite 320, Pasadena, California
  - University of California, San Francisco (UCSF) - Innovation, Technology & Alliances, 1600 Divisadero Street, San Francisco, California
  - UCLA Jonsson Comprehensive Cancer Center, 2020 Santa Monica Boulevard, Santa Monica, California
  - Rocky Mountain Cancer Centers, 1700 South Potomac Street, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion, 1665 Aurora Court, Aurora, Colorado
  - Rocky Mountain Cancer Centers, 4715 Arapahoe Ave, Boulder, Colorado
  - Rocky Mountain Cancer Centers, 2312 N. Nevada Avenue, Suite 400, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, 1800 Williams St., Denver, Colorado
  - Rocky Mountain Cancer Centers, 4700 E. Hale Parkway, Suite 400, Denver, Colorado
  - Rocky Mountain Cancer Centers, 499 E Hampden Ave Suite 450, Englewood, Colorado
  - Rocky Mountain Cancer Centers, 11750 West 2nd Place, Suite 1-100, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, 22 West Dry Creek Circle, Littleton, Colorado
  - Rocky Mountain Cancer Centers, 10103 Ridge Gate Parkway, Suite G-01, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, 2030 W Mountain View Avenue, Ste. 210, Longmont, Colorado
  - Rocky Mountain Cancer Centers, 9397 Crown Crest Blvd., Suite 421, Parker, Colorado
  - Rocky Mountain Cancer Centers, 3676 Parker Blvd., Suite 350, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, 8820 Huron Street, Thornton, Colorado
  - Yale School Of Medicine, New Haven, Connecticut
  - Norwalk Hospital, 34 Maple Street, Norwalk, Connecticut
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute, 601 E. Altamonte Drive, Altamonte Springs, Florida
  - Florida Cancer Specialist, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists & Research Institute, 403 S. King Ave, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists & Research Institute, 3280 McMullen Booth road, Clearwater, Florida
  - Sylvester Comprehensive Cancer Center, Coral Gables, Florida
  - Florida Cancer Specialists & Research Institute, 224 Memorial medical Parway, Daytona Beach, Florida
  - Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, 6420 W Newberry Road Est Wing, Gainesville, Florida
  - Florida Cancer Specialists & Research Institute, 100 Highland Avenue, Largo, Florida
  - Florida Cancer Specialists & Research Institute, 521 N. Lecanto Highway, Lecanto, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists & Research Institute, 8763 River Crossing Blvd, New Port Richey, Florida
  - Florida Cancer Specialists & Research Institute, 1630 SE 18th ST, Ocala, Florida
  - Florida Cancer Specialists & Research Institute, 765 Image Way, Orange City, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Florida Cancer Specialists & Research Institute, 70 W Gore Street, Orlando, Florida
  - Florida Cancer Specialists & Research Institute - 325 Clyde Morris, Ormond Beach, Florida
  - Sylvester Comprehensive Cancer Center, Plantation, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists & Research Institute, 7154 Medical Center Drive, Spring Hill, Florida
  - Florida Cancer Specialists & Research Institute, 1201 Fifth Avenue North, St. Petersburg, Florida
  - Florida Cancer Specialists & Research Institute, 560 Jackson St, St. Petersburg, Florida
  - Florida Cancer Specialists & Research Institute, 3402 W Dr. Martin Luther King Jr Boulevard, Tampa, Florida
  - Florida Cancer Specialists & Research Institute, 4100 Waterman Way, Tavares, Florida
  - Florida Cancer Specialists & Research Institute, 1400 US highway 441 N, The Villages, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Florida Cancer Specialists & Research Institute - 3730 7th Terrace, Vero Beach, Florida
  - Florida Cancer Specialists & Research Institute, 1037 State Road 7 Bldg B, Wellington, Florida
  - Florida Cancer Specialists & Research Institute1309 N Flagler Dr, West Palm Beach, Florida
  - Florida Cancer Specialists & Research Institute, 2100 Glenwood Drive, Winter Park, Florida
  - Atlanta Cancer Center - Alpharetta, Alpharetta, Georgia
  - University Cancer & Blood Center, 3320 Old Jefferson Rd, Athens, Georgia
  - GCS/Annex, Atlanta, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - GCS/Canton, Canton, Georgia
  - Atlanta Cancer Care - Conyers, Conyers, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Atlanta Cancer Care - Decatur, Decatur, Georgia
  - GCS/Stemmer, Decatur, Georgia
  - Atlanta Cancer Care - Stockbridge, Jonesboro, Georgia
  - GCS/Macon, Macon, Georgia
  - GCS/Kennestone, Marietta, Georgia
  - GCS/Northside, Sandy Springs, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Chicago Medical Center 5841 S. Maryland Ave, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital 1900 Silver Cross Blvd, New Lenox, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Orland Park - UCMC Center for Advanced Care 14290 South LaGrange Rd, Orland Park, Illinois
  - MidAmerica Division Inc. c/o Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center - The Richard and Annette Bloch Cancer Care Pavilion, Westwood, Kansas
  - Maryland Oncology Hematology, Bethesda, Maryland
  - Maryland Oncology Hematology, Brandywine, Maryland
  - Maryland Oncology Hematology, Clinton, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Mass General - North Shore Cancer Center ( NSCC ), Danvers, Massachusetts
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology P.A., Coon Rapids, Minnesota
  - Suburban Imaging Northwest, Coon Rapids, Minnesota
  - Suburban Imaging, Coon Rapids, Minnesota
  - Mercy Hospital - Unity Campus AHL, Fridley, Minnesota
  - Minnesota Oncology Hematology P.A., Fridley, Minnesota
  - Minnesota Oncology Hematology P.A., Minneapolis, Minnesota
  - Abbot Northwestern Hospital, Minneapolis, Minnesota
  - Virginia G. Piper Cancer Center at HonorHealth, Minneapolis, Minnesota
  - Mayo Clinic - 200 First Street SW, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, Creve Coeur, Missouri
  - MidAmerica Division Inc. c/o Menorah Medical Center, Independence, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Nebraska Cancer Specialists - Midwest Cancer Center - Papillion, Omaha, Nebraska
  - Nebraska Cancer Specialists - Midwest Cancer Center - Paillion, Omaha, Nebraska
  - Nebraska Cancer Specialists- Midwest Cancer Center- Papillion, Papillion, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - North Shore Hematology Oncology Associates., PC, 235 North Belle Mead Road, East Setauket, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - North Shore Hematology Oncology Associates., PC, 285 Sills Road Building 16, Patchogue, New York
  - UNC Health Care System, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center, 460 W 10th Ave, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, 1145 Olentangy River Road, Columbus, Ohio
  - Providence Medical Group, Portland, Oregon
  - UPMC Hillman Cancer Center Mountainview Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center UPMC East, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center Upper Saint Clair, Pittsburgh, Pennsylvania
  - Allegheny-Singer Research Institute, 320 East North Avenue, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center UPMC Passavant, Pittsburgh, Pennsylvania
  - Tennessee Oncology - Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - Tennesee Oncology - PLLC, Chattanooga, Tennessee
  - Tenesse Oncology - PLLC, Cleveland, Tennessee
  - Tennessee Oncology, LLC, Dickson, Tennessee
  - Tennessee Ocology, LLC, Franklin, Tennessee
  - Tennessee Oncology, LLC, Gallatin, Tennessee
  - West Cancer Center, 7945 Wolf River Blvd, Germantown, Tennessee
  - Tennessee Oncology, LLC, Hermitage, Tennessee
  - Tennessee Oncology, LLC, Lebanon, Tennessee
  - Tennessee Oncology, LLC, Murfreesboro, Tennessee
  - Sarah Cannon Cancer Institute/Tennessee Oncology, Nashville, Tennessee
  - Tennessee Oncology, LLC, Nashville, Tennessee
  - Vanderbilt Breast Cancer Center at One Hundred Oaks 719 Thompson Lane, Suite 25000, Nashville, Tennessee
  - Tennessee Ocology, LLC, Nashville, Tennessee
  - Tenessee Oncology, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic 1301 Medical Center Drive 1903 The Vanderbilt Clinic Nashville, TN 37232, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Tennessee Oncology, LLC, Shelbyville, Tennessee
  - Center for Cancer and Blood Disorders, Arlington, Texas
  - Center for Cancer and Blood Disorders, Burleson, Texas
  - Texas Oncology- Medical City Dallas Building D, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, Denton, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Houston Methodist Hospital - 6565 Fannin St, Houston, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology, Plano, Texas
  - US Oncology, Tyler, Texas
  - Center for Cancer and Blood Disorders, Weatherford, Texas
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Low Moor, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, P.C., Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Cancer Specialists, PC, Woodbridge, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Wytheville, Virginia
  - Swedish Cancer Institute, Edmonds, Washington
  - Swedish Cancer Institute, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Universitair Zlekenhuis Brussel, Brussels
  - UZ Leuven, Leuven
  - Clinique et Maternite Sainte-Elisabeth, Namur
- Canada (5):
  - Cross Cancer Institute, 11560 University Avenue, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, 3755 Côte-Sainte-Catherine, Montreal, Quebec
  - Jewish General Hospital, 3755 Côte-Sainte-Catherine, Québec, Quebec
- France (9):
  - Centre de Lutte Contre le Cancer - Institut de Cancerologie de l'Ouest - Paul Papin, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Florence Lerebours, Saint-Cloud
  - CHU de Nantes - Hôpital Nord Laennec, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (5):
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt
  - Praxis für interdisziplinäre Onkologie & Hämatologie GbR, Freiburg im Breisgau
  - Facharztzentrum Eppendorf, Hamburg
  - Institut für Versorgungsforschung in der Onkologie, Koblenz
  - Praxis für Hämatologie und Internistische Onkologie, Velbert
- Spain (11):
  - Hospital Teresa Herrera, As Xubias, 84, A Coruña
  - Hospital Quirón Barcelona, Plaza Alfonso Comín 5, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Carrer del Mas Casanovas, 90, Barcelona
  - Institut Catala d'Oncologia Hospitalet, Avenida Gran Via 199-203, L'Hospitalet de Llobregat
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complexo Hospitalario Universitario de Santiago (CHUS) - Hospital Clinco Universaitario, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (11):
  - Colchester Hospital University NHS Foundation Trust - Colchester General Hospital, Turner Road, Colchester, ESS
  - The Arden Cancer Centre- University Hospital Coventry, Coventry
  - County Durham and Darlington NHS Foundation Trust - University Hospital of North Durham, Durham
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - The County Hospital, Wye Valley NHS Trust, Hereford
  - The Royal Free London NHS Foundation Trust - The Royal Free Hospital, Pond Street Oncology & Haematology Clinical Trials Unit Dept. of Academic Oncology, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth
  - Taunton and Somerset NHS Foundation Trust - Musgrove Park Hospital, Musgrove Park Hospital, Taunton
  - The Mid Yorkshire Hospitals NHS Trust - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Background] Bardia A, Mayer IA, Vahdat LT, Tolaney SM, Isakoff SJ, Diamond JR, O'Shaughnessy J, Moroose RL, Santin AD, Abramson VG, Shah NC, Rugo HS, Goldenberg DM, Sweidan AM, Iannone R, Washkowitz S, Sharkey RM, Wegener WA, Kalinsky K. Sacituzumab Govitecan-hziy in Refractory Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2019 Feb 21;380(8):741-751. doi: 10.1056/NEJMoa1814213. PMID 30786188
- [Result] Huvitz SA, Tolaney SM, Punie K, et al. 2020 SABCS GS3-06. Biomarker evaluation in the phase 3 ASCENT study of sacituzumab govitecan versus chemotherapy in patients with metastatic triple-negative breast cancer. San Antonio Breast Cancer Symposium; December 8-11, 2020; San Antonio, TX.
- [Result] Dieras V, Weaver R, Tolaney SM, et al. 2020 SABCS PD13-07. Subgroup analysis of patients with brain metastases from the phase 3 ASCENT study of sacituzumab govitecan versus chemotherapy in metastatic triple-negative breast cancer. San Antonio Breast Cancer Symposium; December 8-11, 2020; San Antonio, TX.
- [Result] Rugo HS, Tolaney SM, Loirat D, et al. 2020 SABCS PS11-09. Impact of UGT1A1 status on the safety profile of sacituzumab govitecan in the phase 3 ASCENT study in patients with metastatic triple-negative breast cancer. San Antonio Breast Cancer Symposium; December 8-11, 2020; San Antonio, TX.
- [Result] Bardia A, Tolaney SM, Loirat D, et al. ASCENT: A randomized phase III study of sacituzumab govitecan (SG) vs treatment of physician's choice (TPC) in patients (pts) with previously treated metastatic triple-negative breast cancer (mTNBC). Annals of Oncology (2020) 31 (suppl_4): S1142-S1215. 10.1016/annonc/annonc325
- [Result] Bardia A, Rugo RS, Horne H, et al. A phase III, randomized trial of sacituzumab govitecan (IMMU-132) vs treatment of physician choice (TPC) for metastatic triple-negative breast cancer (mTNBC). Cancer Res. 2018;78 (4 Supplement): OT2-07-05
- [Derived] Loibl S, Loirat D, Tolaney SM, Punie K, Dieras V, Carey LA, Gianni L, Shah A, Phan S, Shi L, Spears PA, Piccart MJ. Summary of quality of life in the ASCENT phase 3 clinical trial for people with metastatic triple-negative breast cancer. Future Oncol. 2024;20(34):2609-2616. doi: 10.1080/14796694.2024.2381408. Epub 2024 Sep 26. PMID 39324726
- [Derived] Hurvitz SA, Bardia A, Punie K, Kalinsky K, Carey LA, Rugo HS, Dieras V, Phan S, Delaney R, Zhu Y, Tolaney SM. Subgroup analyses from the phase 3 ASCENT study of sacituzumab govitecan in metastatic triple-negative breast cancer. NPJ Breast Cancer. 2024 Apr 25;10(1):33. doi: 10.1038/s41523-024-00635-5. PMID 38664404
- [Derived] Bardia A, Rugo HS, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Kalinsky K, Cortes J, Shaughnessy JO, Dieras V, Carey LA, Gianni L, Piccart-Gebhart M, Loibl S, Yoon OK, Pan Y, Hofsess S, Phan SC, Hurvitz SA. Final Results From the Randomized Phase III ASCENT Clinical Trial in Metastatic Triple-Negative Breast Cancer and Association of Outcomes by Human Epidermal Growth Factor Receptor 2 and Trophoblast Cell Surface Antigen 2 Expression. J Clin Oncol. 2024 May 20;42(15):1738-1744. doi: 10.1200/JCO.23.01409. Epub 2024 Feb 29. PMID 38422473
- [Derived] O'Shaughnessy J, Brufsky A, Rugo HS, Tolaney SM, Punie K, Sardesai S, Hamilton E, Loirat D, Traina T, Leon-Ferre R, Hurvitz SA, Kalinsky K, Bardia A, Henry S, Mayer I, Zhu Y, Phan S, Cortes J. Analysis of patients without and with an initial triple-negative breast cancer diagnosis in the phase 3 randomized ASCENT study of sacituzumab govitecan in metastatic triple-negative breast cancer. Breast Cancer Res Treat. 2022 Sep;195(2):127-139. doi: 10.1007/s10549-022-06602-7. Epub 2022 May 11. PMID 35545724
- [Derived] Bardia A, Hurvitz SA, Rugo HS, Brufsky A, Cortes J, Loibl S, Piccart M, Cowden J, Spears P, Carey LA. A plain language summary of the ASCENT study: Sacituzumab Govitecan for metastatic triple-negative breast cancer. Future Oncol. 2021 Oct 1;17(30):3911-3924. doi: 10.2217/fon-2021-0868. Epub 2021 Sep 1. PMID 34467774
- [Derived] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Derived] McCann KE, Hurvitz SA. Innovations in targeted therapies for triple negative breast cancer. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):34-47. doi: 10.1097/GCO.0000000000000671. PMID 33093337
- [Derived] Seligson JM, Patron AM, Berger MJ, Harvey RD, Seligson ND. Sacituzumab Govitecan-hziy: An Antibody-Drug Conjugate for the Treatment of Refractory, Metastatic, Triple-Negative Breast Cancer. Ann Pharmacother. 2021 Jul;55(7):921-931. doi: 10.1177/1060028020966548. Epub 2020 Oct 17. PMID 33070624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Belgium, Canada, France, Germany, Spain, the United Kingdom, and the United States. The first participant was screened on 07 November 2017. The last study visit occurred on 08 December 2020.
Pre-assignment Details: 730 participants were screened.
Groups:
- Sacituzumab Govitecan: Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow intravenous (IV) infusion either by gravity or with an infusion pump on Days 1 and 8 of a 21-day treatment cycle for up to 29.6 months. Infusion rate for the first 15 minutes started with 50 mg/hour or less with a subsequent infusion of 100 to 200 mg/hour up to a maximum recommended rate (advanced every 15 to 30 minutes) of 500 mg/hour with a subsequent infusion of 1000 mg/hour. Participants continued treatment until progression of disease requiring treatment discontinuation or occurrence of unacceptable adverse events (AEs).
- Treatment of Physician's Choice (TPC): Participants received TPC (ie, eribulin, capecitabine, gemcitabine, or vinorelbine), administered as a single-agent regimen that was selected by the investigator before participant randomization. Participants continued treatment until progression of disease requiring treatment discontinuation or occurrence of unacceptable AEs.
  Eribulin was administered IV over 2 to 5 minutes at a dose 1.4 mg/m^2 at North American sites and 1.23 mg/m^2 at European sites on Days 1 and 8 of a 21-day cycle for up to 15.3 months. Lower doses were administered on the same schedule to participants with moderate hepatic impairment (ie, Child-Pugh B; 0.7 mg/m^2 and 0.67 mg/m^2 for North American and European sites, respectively).
  Capecitabine 1000 to 1250 mg/m^2 was administered in a 21-day cycle, with capecitabine administered orally twice daily for 2 weeks followed by 1-week rest period for up to 10.6 months.
  Gemcitabine 800 to 1200 mg/m^2 was administered IV over 30 minutes on Days 1, 8, and 15 of a 28-day cycle for up to 8.1 months.
  Vinorelbine 25 mg/m^2 was administered as a weekly IV injection over 6-10 minutes for up to 11.5 months. Vinorelbine was not allowed as TPC for any participant with Grade 2 neuropathy.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Started | 267 | 262
Enrolled and Treated | 258 | 224
Completed | 0 | 0
Not Completed | 267 | 262
Not completed — Death | 197 | 210
Not completed — Withdrawal of Consent | 11 | 28
Not completed — Lost to Follow-up | 4 | 4
Not completed — Sponsor's Decision | 55 | 20

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population included all randomized participants.
Groups:
- Sacituzumab Govitecan: Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow IV infusion either by gravity or with an infusion pump on Days 1 and 8 of a 21-day treatment cycle for up to 29.6 months. Infusion rate for the first 15 minutes started with 50 mg/hour or less with a subsequent infusion of 100 to 200 mg/hour up to a maximum recommended rate (advanced every 15 to 30 minutes) of 500 mg/hour with a subsequent infusion of 1000 mg/hour. Participants continued treatment until progression of disease requiring treatment discontinuation or occurrence of unacceptable AEs.
- Total: Total of all reporting groups
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC) | Total
Number analyzed (Participants) | 267 | 262 | 529
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.34) | 54.0 (11.69) | 54.0 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 262 | 527
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 25 | 45
  Not Hispanic or Latino | 234 | 226 | 460
  Unknown or Not Reported | 13 | 11 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 13 | 9 | 22
  Race: Black | 28 | 34 | 62
  Race: White | 215 | 203 | 418
  Race: Other | 11 | 16 | 27
Region of Enrollment [Number; unit: participants]
  Belgium | 20 | 25 | 45
  Canada | 3 | 2 | 5
  France | 33 | 29 | 62
  Germany | 0 | 2 | 2
  Spain | 32 | 26 | 58
  United Kingdom | 7 | 8 | 15
  United States | 172 | 170 | 342

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Independent Review Committee (IRC) Assessment in Brain Metastasis Negative (BM-ve) Population
Description: PFS was defined as the time from randomization until objective tumor progression by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death, whichever came first. The date of progression was date of the last observation or radiological assessment of target lesions that either showed a predefined increase (greater than or equal to [≥] 20%) in the sum of the target lesions or the appearance of new non-target lesions. PFS was estimated using Kaplan-Meier estimate.
Time Frame: From randomization until objective tumor progression or death (assessed every 6 weeks for 9 months and then every 9 weeks thereafter until the occurrence of progression of disease; maximum exposure: 29.6 months)
Population: The BM-ve Population included all randomized participants who were randomized to the strata of no baseline brain metastasis at the time of randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
months | 5.6 [4.3 to 6.3] | 1.7 [1.5 to 2.6]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p < 0.0001, Log Rank — Stratified log-rank test and stratified Cox regression adjusted for stratification factors: number of prior chemotherapies, presence of known brain metastases at study entry, and region; Hazard Ratio (HR) = 0.387, 95% CI 2-sided [0.305 to 0.492]

2. Secondary Outcome: Progression-Free Survival (PFS) by IRC Assessment in the ITT Population
Description: PFS was defined as the time from randomization until objective tumor progression by RECIST v1.1 or death, whichever came first. The date of progression was date of the last observation or radiological assessment of target lesions that either showed a predefined increase (≥20%) in the sum of the target lesions or the appearance of new non-target lesions. PFS was estimated using Kaplan-Meier estimate.
Time Frame: as for outcome 1
Population: The ITT Population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 267 | 262
months | 4.8 [4.1 to 5.8] | 1.7 [1.5 to 2.5]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.413, 95% CI 2-sided [0.330 to 0.517]

3. Secondary Outcome: Overall Survival (OS) in BM-ve Population
Description: Overall survival (OS) was defined as the time from the randomization to death from any cause. OS was estimated using Kaplan-Meier estimate.
Time Frame: From the randomization to death from any cause (maximum follow-up duration: 30.8 months)
Population: Participants in the BM-ve Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
months | 12.1 [10.7 to 14.0] | 6.7 [5.8 to 7.7]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p < 0.0001, Log Rank — Stratified log-rank test and stratified Cox regression adjusted for stratification factors: number of prior chemotherapies and region; Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.390 to 0.592]

4. Secondary Outcome: Overall Survival (OS) in ITT Population
Description: as for outcome 3
Time Frame: From the randomization to death from any cause (maximum follow-up duration: 30.8 months)
Population: Participants in the ITT Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 267 | 262
months | 11.8 [10.5 to 13.8] | 6.9 [5.9 to 7.7]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.514, 95% CI 2-sided [0.422 to 0.625]

5. Secondary Outcome: Objective Response Rate (ORR) by IRC and Investigator Assessment in BM-ve Population
Description: ORR was defined as the percentage of participants who had the overall best response as either a confirmed complete response (CR) or partial response (PR) relative to the size of population under evaluation. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; and no new lesions. PR: ≥30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; and no new lesions.
Time Frame: From randomization to the date of progression or death (assessed every 6 weeks for 9 months and then every 9 weeks thereafter until the occurrence of progression of disease; maximum exposure: 29.6 months)
Population: Participants in the BM-ve Population with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
percentage of participants
  ORR by IRC Assessment: number analyzed (Participants) | 230 | 230
  ORR by IRC Assessment | 34.9 [28.8 to 41.4] | 4.7 [2.4 to 8.3]
  ORR by Investigator Assessment | 33.2 [27.2 to 39.6] | 6.4 [3.6 to 10.4]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); ORR by IRC Assessment; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 10.859, 95% CI 2-sided [5.590 to 21.095]
Statistical Analysis 2: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); ORR by Investigator Assessment; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7.363, 95% CI 2-sided [4.063 to 13.341]

6. Secondary Outcome: Time to Objective Response by the Investigator Assessment in BM-ve Population
Description: Time to response was defined as the time from randomization to the first recorded objective response (ie, CR or PR). CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; and no new lesions. PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; and no new lesions.
Time Frame: From randomization to the first recorded objective response (assessed every 6 weeks for 9 months and then every 9 weeks thereafter until the occurrence of progression of disease; maximum exposure: 29.6 months)
Population: Participants in the BM-ve Population with objective response were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 78 | 15
months | 2.14 (1.322) | 2.72 (2.933)

7. Secondary Outcome: Time to Objective Response by the IRC Assessment in BM-ve Population
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Participants in the BM-ve Population with objective response were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 82 | 11
months | 2.67 (1.913) | 1.86 (0.919)

8. Secondary Outcome: Duration of Response (DOR) by IRC and Investigator Assessment in BM-ve Population
Description: DOR was defined as the number of days between the first date showing a documented response of CR or PR and the date of progression or death. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; and no new lesions. PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; and no new lesions. The date of progression was date of the last observation or radiological assessment of target lesions that either showed a predefined increase (≥20%) in the sum of the target lesions or the appearance of new non-target lesions.
Time Frame: From the first date of documented response of CR or PR to the date of progression or death (assessed every 6 weeks for 9 months and then every 9 weeks thereafter until the occurrence of progression of disease; maximum exposure: 29.6 months)
Population: Participants in the BM-ve Population with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 82 | 15
months
  IRC Assessment: number analyzed (Participants) | 82 | 11
  IRC Assessment | 6.3 [5.5 to 7.9] | 3.6 [2.8 to NA] — Due to smaller number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated.
  Investigator Assessment: number analyzed (Participants) | 78 | 15
  Investigator Assessment | 6.9 [5.6 to 7.9] | 3.0 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); DOR by IRC Assessment; Test type: Other; p = 0.0683, Log Rank — Stratified log-rank test and stratified Cox regression adjusted for stratification factors: number of prior chemotherapies, and region; Hazard Ratio (HR) = 0.407, 95% CI 2-sided [0.150 to 1.107]
Statistical Analysis 2: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); DOR by Investigator Assessment; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 8, analysis 1]; Hazard Ratio (HR) = 0.212, 95% CI 2-sided [0.103 to 0.435]

9. Secondary Outcome: Time to Progression (TTP) by Investigator Assessment in BM-ve Population
Description: Time to Progression (TTP) was defined as the time from the date of randomization to the date of the first evidence of disease progression as assessed using RECIST 1.1 criteria. The date of progression was date of the last observation or radiological assessment of target lesions that either showed a predefined increase (≥20%) in the sum of the target lesions or the appearance of new non-target lesions. Participants without progression were censored.
Time Frame: From randomization until disease progression (assessed every 6 weeks for 9 months and then every 9 weeks thereafter until the occurrence of progression of disease; maximum exposure: 29.6 months)
Population: Participants in the BM-ve Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
months | 5.7 [5.2 to 6.9] | 1.8 [1.5 to 2.6]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); TTP by Investigator Assessment; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.317, 95% CI 2-sided [0.248 to 0.404]

10. Secondary Outcome: Time to Progression (TTP) by IRC Assessment in BM-ve Population
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Participants in the BM-ve Population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
months | 5.8 [4.8 to 6.9] | 2.1 [1.5 to 2.7]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); TTP by IRC Assessment; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.406, 95% CI 2-sided [0.315 to 0.525]

11. Secondary Outcome: Clinical Benefit Rate (CBR) by IRC and Investigator Assessment in BM-ve Population
Description: CBR was defined as the percentage of participants with best response as either CR, PR, or stable disease (SD) with a duration of ≥6 months. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; and no new lesions. PR: ≥30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; and no new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started; and Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits. PD: ≥20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since treatment started or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 5
Population: Participants in the BM-ve Population were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 235 | 233
percentage of participants
  IRC Assessment | 44.7 [38.2 to 51.3] | 8.6 [5.3 to 12.9]
  Investigator Assessment | 45.5 [39.0 to 52.1] | 10.3 [6.7 to 14.9]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); CBR by IRC Assessment; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 8.543, 95% CI 2-sided [5.055 to 14.437]
Statistical Analysis 2: Comparison: Sacituzumab Govitecan vs Treatment of Physician's Choice (TPC); CBR by Investigator Assessment; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7.492, 95% CI 2-sided [4.540 to 12.364]

12. Secondary Outcome: Percentage of Participants Experiencing Any Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and TEAEs Leading to Discontinuation of Study Drug
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 4.03. An AE that met one or more of the following outcomes was classified as serious:
  * Fatal
  * Life-threatening
  * Disabling/incapacitating
  * Results in hospitalization or prolongs a hospital stay
  * A congenital abnormality
  * Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: First dose date up to last follow-up (maximum up to 30.8 months)
Population: Safety Population included all participants who received at least one dose of sacituzumab govitecan or TPC.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 258 | 224
percentage of participants
  Any TEAEs | 99.6 | 97.8
  SAEs | 26.7 | 28.6
  TEAEs Leading to Discontinuation of Study Drug | 4.7 | 5.4

13. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ-C30) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess quality of life (QoL), it is composed of 30 questions (items) resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, pain), and 6 single items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status indicate a better quality of life; a positive change from baseline indicates improvement. Lower scores on the symptom and single-item scales indicate a better quality of life; a negative change from baseline indicates improvement.
Time Frame: Baseline; End of Treatment (EOT) (up to 29.6 months)
Population: Participants in the Safety analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 258 | 224
score on a scale
  Global Health Status/QoL: Baseline: number analyzed (Participants) | 247 | 217
  Global Health Status/QoL: Baseline | 61.9 (21.31) | 56.4 (22.21)
  Global Health Status/QoL: Change From Baseline at EOT: number analyzed (Participants) | 181 | 147
  Global Health Status/QoL: Change From Baseline at EOT | -5.8 (22.71) | -9.4 (20.46)
  Physical Functioning: Baseline: number analyzed (Participants) | 248 | 217
  Physical Functioning: Baseline | 73.2 (21.69) | 71.2 (21.24)
  Physical Functioning: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Physical Functioning: Change From Baseline at EOT | -4.6 (21.07) | -13.5 (20.54)
  Role Functioning: Baseline: number analyzed (Participants) | 248 | 217
  Role Functioning: Baseline | 68.1 (30.35) | 65.1 (30.31)
  Role Functioning: Change From Baseline at EOT: number analyzed (Participants) | 183 | 146
  Role Functioning: Change From Baseline at EOT | -8.4 (32.87) | -18.8 (29.83)
  Emotional Functioning: Baseline: number analyzed (Participants) | 247 | 217
  Emotional Functioning: Baseline | 71.9 (22.33) | 68.9 (23.87)
  Emotional Functioning: Change From Baseline at EOT: number analyzed (Participants) | 182 | 147
  Emotional Functioning: Change From Baseline at EOT | -3.8 (25.02) | -3.5 (22.16)
  Cognitive Functioning: Baseline: number analyzed (Participants) | 247 | 217
  Cognitive Functioning: Baseline | 81.7 (21.08) | 79.5 (23.91)
  Cognitive Functioning: Change From Baseline at EOT: number analyzed (Participants) | 182 | 147
  Cognitive Functioning: Change From Baseline at EOT | -7.5 (22.81) | -6.1 (22.92)
  Social Functioning: Baseline: number analyzed (Participants) | 247 | 216
  Social Functioning: Baseline | 69.1 (29.96) | 69.6 (26.88)
  Social Functioning: Change From Baseline at EOT: number analyzed (Participants) | 182 | 145
  Social Functioning: Change From Baseline at EOT | -5.9 (27.52) | -10.3 (29.60)
  Fatigue: Baseline: number analyzed (Participants) | 248 | 217
  Fatigue: Baseline | 39.4 (25.72) | 42.1 (25.99)
  Fatigue: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Fatigue: Change From Baseline at EOT | 5.1 (25.93) | 14.0 (23.05)
  Nausea and Vomiting: Baseline: number analyzed (Participants) | 248 | 217
  Nausea and Vomiting: Baseline | 8.3 (16.36) | 10.3 (18.26)
  Nausea and Vomiting: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Nausea and Vomiting: Change From Baseline at EOT | 5.2 (23.93) | 7.3 (23.33)
  Pain: Baseline: number analyzed (Participants) | 248 | 217
  Pain: Baseline | 37.9 (30.54) | 42.5 (30.38)
  Pain: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Pain: Change From Baseline at EOT | 2.8 (27.84) | 6.8 (30.33)
  Dyspnoea: Baseline: number analyzed (Participants) | 248 | 217
  Dyspnoea: Baseline | 25.4 (30.36) | 25.0 (29.09)
  Dyspnoea: Change From Baseline at EOT: number analyzed (Participants) | 180 | 146
  Dyspnoea: Change From Baseline at EOT | 0.7 (30.91) | 5.9 (28.95)
  Insomnia: Baseline: number analyzed (Participants) | 248 | 217
  Insomnia: Baseline | 33.2 (30.95) | 35.6 (31.42)
  Insomnia: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Insomnia: Change From Baseline at EOT | 4.4 (34.67) | -4.3 (32.24)
  Appetite Loss: Baseline: number analyzed (Participants) | 248 | 217
  Appetite Loss: Baseline | 20.8 (27.34) | 25.8 (28.68)
  Appetite Loss: Change From Baseline at EOT: number analyzed (Participants) | 183 | 147
  Appetite Loss: Change From Baseline at EOT | 3.1 (31.78) | 10.0 (30.32)
  Constipation: Baseline: number analyzed (Participants) | 247 | 217
  Constipation: Baseline | 17.7 (27.18) | 19.0 (26.56)
  Constipation: Change From Baseline at EOT: number analyzed (Participants) | 182 | 147
  Constipation: Change From Baseline at EOT | 3.3 (28.92) | 7.0 (31.27)
  Diarrhoea: Baseline: number analyzed (Participants) | 247 | 217
  Diarrhoea: Baseline | 7.2 (17.73) | 6.5 (15.69)
  Diarrhoea: Change From Baseline at EOT: number analyzed (Participants) | 182 | 147
  Diarrhoea: Change From Baseline at EOT | 11.4 (28.56) | 3.6 (22.46)
  Financial Difficulties: Baseline: number analyzed (Participants) | 246 | 217
  Financial Difficulties: Baseline | 27.6 (34.39) | 22.4 (30.91)
  Financial Difficulties: Change From Baseline at EOT: number analyzed (Participants) | 181 | 147
  Financial Difficulties: Change From Baseline at EOT | 0.4 (24.09) | 1.1 (23.54)

14. Secondary Outcome: Percentage of Participants Experiencing the Worst Laboratory Abnormalities Grade 3 or 4 Post-Baseline
Description: Blood samples were collected for hematology, serum chemistry and the laboratory abnormalities were assessed. The most severe graded abnormality observed post-baseline for each graded test was counted for each participant. Safety as assessed by grading of laboratory values and AEs according to the National Cancer Institutes' Common Terminology Criteria for Adverse Events (NCI CTCAE) covering grades 0-5 (0=Normal, 1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening, 5=Death). The percentage of participants with worst postbaseline grades 3 or 4 are reported.
Time Frame: First dose date up to last follow-up (maximum up to 30.8 months)
Population: Participants in the Safety analysis set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
Number analyzed (Participants) | 258 | 224
percentage of participants
  Anemia | 8.9 | 5.4
  Lymphocyte Count Decreased | 33.3 | 25.0
  Neutrophil Count Decreased | 48.8 | 35.3
  Platelet Count Decreased | 1.2 | 2.7
  White Blood Cell Decreased | 41.1 | 25.4
  Alanine Aminotransferase Increased | 1.2 | 2.2
  Alkaline Phosphatase Increased | 3.1 | 3.6
  Aspartate Aminotransferase Increased | 3.5 | 2.2
  Blood Bilirubin Increased | 1.9 | 2.7
  Creatinine Increased | 0.4 | 0
  Hypercalcemia | 0 | 0.4
  Hyperglycemia | 3.1 | 3.1
  Hyperkalemia | 0.8 | 0
  Hypermagnesemia | 0.4 | 0.4
  Hypernatremia | 0 | 0
  Hypoalbumenemia | 0.8 | 1.3
  Hypocalcemia | 1.6 | 1.3
  Hypoglycemia | 0.4 | 0
  Hypokalemia | 4.3 | 0.9
  Hypomagnesemia | 0.8 | 0
  Hyponatremia | 3.9 | 3.6
  Hypophosphatemia | 8.1 | 3.6

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last follow-up (maximum up to 30.8 months); All-Cause Mortality: From randomization up to 30.8 months
Description: Serious Adverse Events and Other Adverse Events: Safety Population included all participants who received at least one dose of sacituzumab govitecan or TPC.
  All-Cause Mortality: The ITT Population included all randomized participants.
Arm/Group | Sacituzumab Govitecan | Treatment of Physician's Choice (TPC)
All-Cause Mortality (participants affected / at risk) | 201/267 | 222/262
Serious Adverse Events (participants affected / at risk) | 69/258 | 64/224
Other Adverse Events (participants affected / at risk) | 256/258 | 213/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (N=258) | Treatment of Physician's Choice (TPC) (N=224)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 5
Swelling (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 2
Corynebacterium infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 4
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Breast ulceration (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (N=258) | Treatment of Physician's Choice (TPC) (N=224)
Anaemia (Blood and lymphatic system disorders) | 102 | 61
Neutropenia (Blood and lymphatic system disorders) | 108 | 56
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 14
Abdominal pain (Gastrointestinal disorders) | 54 | 16
Abdominal pain upper (Gastrointestinal disorders) | 23 | 8
Constipation (Gastrointestinal disorders) | 96 | 52
Diarrhoea (Gastrointestinal disorders) | 168 | 38
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 7
Nausea (Gastrointestinal disorders) | 160 | 68
Stomatitis (Gastrointestinal disorders) | 27 | 14
Vomiting (Gastrointestinal disorders) | 85 | 36
Asthenia (General disorders) | 39 | 28
Chills (General disorders) | 14 | 6
Fatigue (General disorders) | 133 | 89
Mucosal inflammation (General disorders) | 20 | 14
Oedema peripheral (General disorders) | 25 | 24
Pain (General disorders) | 18 | 11
Pyrexia (General disorders) | 37 | 27
Nasopharyngitis (Infections and infestations) | 18 | 5
Upper respiratory tract infection (Infections and infestations) | 32 | 7
Urinary tract infection (Infections and infestations) | 35 | 17
Alanine aminotransferase increased (Investigations) | 28 | 22
Aspartate aminotransferase increased (Investigations) | 30 | 27
Blood alkaline phosphatase increased (Investigations) | 17 | 12
Lymphocyte count decreased (Investigations) | 20 | 13
Neutrophil count decreased (Investigations) | 71 | 45
Platelet count decreased (Investigations) | 7 | 15
Weight decreased (Investigations) | 22 | 15
White blood cell count decreased (Investigations) | 33 | 23
Decreased appetite (Metabolism and nutrition disorders) | 71 | 46
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 17 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 46 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 32 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 15 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 17
Dizziness (Nervous system disorders) | 28 | 16
Dysgeusia (Nervous system disorders) | 22 | 6
Headache (Nervous system disorders) | 47 | 28
Neuropathy peripheral (Nervous system disorders) | 9 | 24
Anxiety (Psychiatric disorders) | 17 | 8
Insomnia (Psychiatric disorders) | 30 | 11
Breast pain (Reproductive system and breast disorders) | 14 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 61 | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 41
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 121 | 36
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 7
Rash (Skin and subcutaneous tissue disorders) | 32 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 3
Hypertension (Vascular disorders) | 17 | 14
Lymphoedema (Vascular disorders) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After study conclusion and without prior written approval from Immunomedics and Gilead sciences, investigators in this study may communicate, orally present/publish in scientific journals/other media only after following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Immunomedics and Gilead sciences in an abstract, manuscript/presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02574455/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT02574455/SAP_002.pdf